CLINICAL TRIAL: NCT00806429
Title: Transvaginal Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0712003306
Record Dates: First submitted 2008-12-02; First posted 2008-12-10 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2012-01

CONDITIONS: Appendicitis
Keywords: appendicitis; surgery; laparoscopy; natural orifice transluminal surgery
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): transvaginal appendectomy
  Interventions: Procedure: transvaginal appendectomy
- 2 (No Intervention)

INTERVENTIONS:
Procedure: transvaginal appendectomy — patient undergoes transvaginal appendectomy
  Arms: 1

SUMMARY:
The purpose of this study is to determine the feasibility and safety of transvaginal appendectomy and determine and compare the postoperative pain and quality of life after surgery to standard laparoscopic transabdominal appendectomy.

ELIGIBILITY:
Inclusion Criteria:

* ultrasound or CT-based diagnosis of acute or chronic appendicitis
* ASA classification 1 or 2

Exclusion Criteria:

* BMI >35
* on Immunosuppressive meds or immunocompromised
* on blood thinners or aspirin or abnormal coagulation tests
* h/o ectopic pregnancy, PID or endometriosis
* prior open abdominal surgery or transvaginal surgery
* with diffuse peritonitis
* evidence of abscess
* retroflexed uterus
* non english speaking

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
feasibility of transvaginal appendectomy | 1 year

SECONDARY OUTCOMES:
pain | 1 year
quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E Roberts, MD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Roberts KE, Solomon D, Mirensky T, Silasi DA, Duffy AJ, Rutherford T, Longo WE, Bell RL. Pure transvaginal appendectomy versus traditional laparoscopic appendectomy for acute appendicitis: a prospective cohort study. Ann Surg. 2012 Feb;255(2):266-9. doi: 10.1097/SLA.0b013e31823b2748. PMID 22167005